CLINICAL TRIAL: NCT05591105
Title: Post-operative Morphine Consumption in Obese Patients Undergoing Laparoscopic Bariatric Surgery Following Ketamina and Lidocaine Perfusion
Brief Title: The Postoperative Lidocaine and Ketamine Effects on Morphine Requirement in Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Tiva Group (Other)
Responsible Party: Principal Investigator, Carolina Frederico, Principal Investigator, Tiva Group
Other Study IDs: TIVA OFA Obese patients
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pharmacological Action; Post Operative Pain; Opioid Use; Obesity, Morbid; Anesthesia Morbidity
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid | interventions — Control Groups; dexketoprofen trometamol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A:: At the end of surgery, on the recovery room, this group will receive lidocaine (1 mg/kg/h) and Ketamine (0,15 mg/kg/h) for 90 minutes
  Interventions: Drug: Control Group
- Group B:: At the end of surgery, on the recovery room, this group will receive placebo (normal salin solution) for 90 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Control Group — At the end of surgery, they will continue receiving analgesia according the schedule and, addicionally, lidocaine (1 mg/kg/h) and Ketamine (0,15 mg/kg/h) for 90 minute as part of postoperative analgesia.
  Other Names: Multimodal analgesia will be performed with paracetamol 1 gr, dexketoprofen 50 mg and metamizol 2 gr and morphine according to visual analogue scale
  Groups: Group A:
Drug: Placebo — At the end of surgery, they will continue receiving analgesia according the schedule.
  Other Names: Multimodal analgesia will be performed with paracetamol 1 gr, dexketoprofen 50 mg and metamizol 2 gr and morphine according to visual analogue scale
  Groups: Group B:

SUMMARY:
The goal of this observational study is to evaluate the quality of postoperative analgesia in a group of obese patients schedule to bariatric surgery under TIVA Opiod-free after to receive lidocaine and ketamine perfusion. The main question it aims to answer are: How lidocaine and ketamine perfusion during recovery period does impact over morphine consumption on the following 48 hours after surgery? All participants will receive total intravenous anesthesia and, at the end of the surgery, they will be divided in two groups, group A: placebo and, group B: with postoperative lidocaine and ketamine perfusion. Our hypothesis is ketamine and lidocaine are a good alternative to decrease the use of morphine in obese patients.

DETAILED DESCRIPTION:
The obese patients have more risk for certain side effects and complications with elevated risk of perioperative mortality and morbidity. An effective postoperative pain management is important to prevent pulmonary complications and, it is not recommended continuous infusions of opioids in this kind of patients, because the opioid-induced upper airway obstruction and respiratory depression are more likely to be seen in obese patients with obstructive sleep apnea. We can reduce perioperative opioid using dexmedetomidine, ketamine and lidocaine, however, it is a little know the use and benefits of lidocaine and ketamine inmediately after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 18 y 65 years old.
* IMC > 30 kg/m2
* ASA II/III

Exclusion Criteria:

* Patients taking high doses of opioids before operation for chronic pain
* Patients with allergies to any study medication.
* Pregnancy or breastfeeding.
* Kidney or heptic failure.
* Surgical complication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patient schedule to laparoscopic bariatric surgery since january 2022 until diciembre 2022 at Hospital HM Delfos Barcelona España.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 48 hours
  The visual analog scale (VAS) will be used to measure pain on recovery room and hospitalization area.

OTHER OUTCOMES:
Kind of surgery | During surgery
  The laparoscopic Sleeve Gastrectomy is technically more simple and shorter surgery time than the Roux-en-Y Gastric Bypass and maybe less painfull

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Frederico, Principal Investigator — Tivagrooup; Gregory Contreras-Pérez, Principal Investigator — Tiva Group
Locations (1):
- Carolina, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No